CLINICAL TRIAL: NCT07000188
Title: Preoperative Ultrasonographic Assesment of the Internal Jugular Vein to Predict Post Spinal Hypotension in Elderly Patients, Observational Study
Brief Title: Jugular Ultrasound for Spinal Hypotension
Acronym: JUSH
Status: Active, not recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai younes Taha, lecturer of anesthesia at cairo university hospital., Cairo University
Other Study IDs: ANES -IJV U/S 2025
Record Dates: First submitted 2025-05-23; First posted 2025-06-02 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hypotension; Anesthesia, Spinal; Aged
Keywords: spinal anesthesia; elderly; hypotension; ultrasound; passive leg raising; IJV
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spinal induced hypotension is common complication in geriatric group of patient with percentage up to 73% among these group]. the most common causes that enhance occurrence of post spinal anesthesia induced hypotension among elderly are poor physical condition , chronic systemic diseases , medications and long fasting time, intraoperative hypotension if severe or prolonged is associated with hazardous complication such as myocardial infarction , stroke, renal failure and perioperative mortality ,so accurate assessment of intravascular volume before induction of anesthesia is necessary to limit these hazards.

Various studies had reported that ultrasonographic measurements of inferior vena cava collapsibility index is a good predictor for reflexing the intravascular volume status[5][6] , this is non invasive , on the other hand IVC is not easily feasible in obese and pregnant women.

Some studies compared the difference between IVC and IJV as predictor marker for fluid responsiveness and reported that right internal jugular vein distensibility appears to be a surrogate marker for inferior vena cava vein distensibility for evaluating fluid responsiveness.

Almost great percentage of anesthesiologist easily use IJV ultrasonography for catheterization and it is easily feasible in almost all patients, recent studies documented that noninvasive ultrasonographic measurements of internal jagular vein diameter has a role in assessment of intravascular volume status in spontaneously and mechanically breathing patients, Passive leg raising has been shown to be useful in assessing intravascular volume depletion or fluid responsiveness , some studies compared IJV changing in diameter for supine and trendelenburg positions, there is a similar change in IJV diameter will occur with passive leg raising positions , trendelenburg position may be disadvantageous as it impair gas function and cardiac function especially in elderly and obese patients , on the other hand passive leg raising is simpler and more comfortable to the elderly.

Finally preoperative detection of decreased intravascular volume is crucial in elderly patients, so we hypothesized that preoperative ultrasonographic evaluation of the internal jagular vein measurements may be a reliable tool for estimating intravascular volume and prediction of post spinal hypotension in elderly.

ELIGIBILITY:
Inclusion Criteria:

* • Age > 65 years old.

  * Both sexes.
  * American Society of Anesthesiologists (ASA) physical status I, II , III.
  * Elective surgeries Under spinal anesthesia in the supine position.

Exclusion Criteria:

* • Body Mass Index (BMI) more than 35 kg/m2.

  * Uncontrolled hypertension.
  * Ejection fraction less than 40%
  * Emergency cases.
  * Absolute or relative contraindications to spinal anesthesia.
  * Patients with a baseline arterial systolic blood pressure (SBP) less than 90 mmHg or mean arterial blood pressure (MBP) less than 65 mmHg.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: elderly patients equal or more than 65 years old
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
• The accuracy of ultrasonographic changes in IJV area with positions (supine and PLR) in predicting spinal hypotension in geriatric patients. | time needed to spinal anesthesia related hypotension occurs which arround 20 to 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt